CLINICAL TRIAL: NCT04654208
Title: Palbociclib Treatment Patterns in Swedish Patients With Metastatic Breast Cancer - Swedish Ibrance Registries Insights (SIRI)
Brief Title: Swedish Ibrance Registries Insights (SIRI)
Acronym: SIRI
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481158; SIRI (Other: Alias Study Number)
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Malignant Neoplasm of Breast
Keywords: metastatic breast cancer (MBC)
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HR+/HER2- locally advanced or MBC in combination with an aromatase inhibitor (AI): Group Description: patients with at least one filled prescription of palbociclib (ATC (anatomic therapeutic chemical classification system ) code: L01XE33)
  Interventions: Drug: palbociclib
- HR+/HER2- locally advanced or MBC cancer in combination with fulvestrant: Group Description: patients with at least one filled prescription of palbociclib ATC (code: L01XE33)
  Interventions: Drug: palbociclib

INTERVENTIONS:
Drug: palbociclib — patients on palbociclib combination treatment

SUMMARY:
The main objectives of this study are to describe patient characteristics, treatment patterns and clinical outcomes of patients receiving palbociclib in Swedish clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. One or more (≥1) filled prescription of palbociclib (ATC code: L01XE33)
2. Age ≥18 years at index date

Exclusion Criteria:

There are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all adult (age ≥18 years) patients (male and female) with at least one filled prescription of palbociclib (ATC code: L01XE33) registered in the Swedish Prescribed Drug Register between January 1st, 2017 and June 30th 2020.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients on treatment | 01 January 2017 until 30 September 2020
  Proportion of patients who have not discontinued treatment will be assessed at various timepoints (Time Frame: treatment start date through end of study [assessed up to 48 months])

SECONDARY OUTCOMES:
Proportion of patients alive | 01 January 2017 until 30 September 2020
  Proportion of patients alive on palbociclib combination treatment at different points in time (Time Frame: treatment start date through end of study [assessed up to 48 months])
Describe the demographic and clinical characteristics of the patient population receiving palbociclib combination treatment | 01 January 2017 until 30 September 2020

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Sweden, Sollentuna, Sweden

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481158